CLINICAL TRIAL: NCT00059852
Title: A Phase II Study of OSI-774 (Tarceva) and Gemcitabine for Patients With Metastatic Breast Cancer
Brief Title: Erlotinib and Gemcitabine in Treating Patients With Metastatic Breast Cancer Previously Treated With An Anthracycline and/or a Taxane
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0234; NCI-2012-02529 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000298778 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: male breast cancer; recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine + erlotinib (Experimental): Patients receive gemcitabine IV on days 1 and 8 and oral erlotinib on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Patients achieving a complete response are followed every 6 weeks for up to 5 years or until disease progression (PD). Patients discontinuing study therapy for any other reason are followed every 3 months until PD and then every 6 months for up to 5 years.
  Interventions: Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as gemcitabine work in different ways to stop tumor cells from dividing so they stop growing or die. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Combining gemcitabine with erlotinib may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine with erlotinib in treating patients who have metastatic breast cancer that has been previously treated with an anthracycline and/or a taxane.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the anti-tumor activity of erlotinib and gemcitabine in patients with metastatic breast cancer previously treated with anthracycline and/or taxane.
* Determine the adverse event profile of this regimen in these patients.
* Determine whether epidermal growth factor receptor and HER-2 receptor intensity and serum concentrations have an impact on clinical response in patients treated with this regimen.
* Determine the impact of genetic differences in proteins involved in drug response (transport, metabolism, and mechanism of action) on clinical response and adverse events associated with gemcitabine in these patients.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV on days 1 and 8 and oral erlotinib on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients achieving a complete response are followed every 6 weeks for up to 5 years or until disease progression (PD). Patients discontinuing study therapy for any other reason are followed every 3 months until PD and then every 6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed breast cancer

  * Clinical evidence of metastatic disease
* Candidate for first- or second-line chemotherapy for metastatic disease
* Must have received prior anthracycline or taxane therapy (may have had both in the neoadjuvant, adjuvant, or metastatic setting)
* At least 1 measurable lesion at least 20 mm by CT scan or MRI OR at least 10 mm by spiral CT scan

  * The following are not considered measurable disease:

    * Small lesions less than 20 mm by CT scan or MRI
    * Bone lesions
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* No active CNS metastases (treated CNS metastases stable for more than 8 weeks are allowed)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8.5 g/dL

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 3 times ULN
* Alkaline phosphatase no greater than 3 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Gastrointestinal

* No inability to take oral or nasogastric medication
* No requirement for IV alimentation
* No active peptic ulcer disease

Ophthalmic

* No abnormalities of the cornea based on history (e.g., dry eye syndrome or Sjögren's syndrome)
* No congenital abnormality (e.g., Fuch's dystrophy)
* No abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
* No abnormal corneal sensitivity test (Schirmer test or similar tear production test)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

  * Sub-dermal implants and condoms are not considered acceptable forms of contraception
* No other invasive non-breast malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 2 weeks since prior immunotherapy
* No prior cetuximab

Chemotherapy

* At least 2 weeks since prior chemotherapy and recovered
* No more than 1 prior chemotherapy regimen for metastatic disease
* No more than 2 prior chemotherapy regimens total, including adjuvant therapy

Endocrine therapy

* Prior hormonal therapy allowed in metastatic and/or adjuvant setting

Radiotherapy

* At least 2 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of bone marrow
* No prior strontium chloride Sr 89

Surgery

* More than 4 weeks since prior major surgery
* No prior surgical procedures affecting absorption

Other

* No prior epidermal growth factor receptor-targeting therapies (e.g., gefitinib or EKB-569)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent antitumor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2003-06; Primary Completion 2006-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 5 years

SECONDARY OUTCOMES:
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Edith A. Perez, MD, Study Chair — Mayo Clinic
Locations (25):
- United States (25):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin

REFERENCES:
- [Background] Reinholz MM, Kitzmann KA, Tenner K, Hillman D, Dueck AC, Hobday TJ, Northfelt DW, Moreno-Aspitia A, Roy V, LaPlant B, Allred JB, Stella PJ, Lingle WL, Perez EA. Cytokeratin-19 and mammaglobin gene expression in circulating tumor cells from metastatic breast cancer patients enrolled in North Central Cancer Treatment Group trials, N0234/336/436/437. Clin Cancer Res. 2011 Nov 15;17(22):7183-93. doi: 10.1158/1078-0432.CCR-11-0981. Epub 2011 Oct 5. PMID 21976532
- [Background] Pockaj BA, Mukherjee P, Tinder TL, et al.: NCCTG N0338: effect of docetaxel and carboplatin on VEGF, PGE2, and immune cells in patients with stage II or III breast cancer. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-5110, 2008.
- [Background] Reinholz MM, Kitzmann KK, Hillman D, et al.: Differential gene expression in circulating tumor cells between primary and metastatic breast cancer patients. [Abstract] Breast Cancer Res Treat 106 (1): A-5022, S213-4, 2007.
- [Result] Thome S, Hobday T, Hillman D, et al.: Translational correlates, including outcome for patients with ER-/PR-/HER2- (triple negative (TNeg)) disease from N0234, a phase II trial of gemcitabine and erlotinib for pts with previously treated metastatic breast cancer (MBC). [Abstract] J Clin Oncol 25 (Suppl 18): A-1071, 2007.
- [Result] Graham DL, Hillman DW, Hobday TJ, et al.: N0234: phase II study of erlotinib (OSI-774) plus gemcitabine as first-or second-line therapy for metastatic breast cancer (MBC). [Abstract] J Clin Oncol 23 (Suppl 16): A-644, 39s, 2005.